CLINICAL TRIAL: NCT01503125
Title: Clinical Study of Giant Axonal Neuropathy
Brief Title: Giant Axonal Neuropathy Natural History Study
Status: Terminated | Type: Observational
Why Stopped: PI left the institution
Sponsor: Columbia University (Other)
Collaborators: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Other Study IDs: AAAI4500
Record Dates: First submitted 2011-12-29; First posted 2012-01-02 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2017-01

CONDITIONS: Giant Axonal Neuropathy
Keywords: GAN; Giant Axonal Neuropathy; Neuromuscular Disease; Natural History Study; Observational Study
MeSH Terms: conditions — Giant Axonal Neuropathy; Neuromuscular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Skin Tissue, Blood, Cerebrospinal fluid (CSF)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Giant Axonal Neuropathy (GAN) is a devastating and rare childhood disease. Children with GAN develop increasing muscle weakness, impaired sensation, and at times mental retardation. GAN starts in infancy, leads to significant disability, and typically leads to death within the first 30 years of life. GAN is caused by a defect in the "gigaxonin" (GAN) gene, resulting in pathologically enlarged and dysfunctional nerves. Currently, there is no effective therapy. To find out what medications can help patients with GAN, the investigators have to conduct clinical trials. In this study, the investigators propose to prepare for future clinical trials and will invite GAN patients to join our research effort.

The investigators will examine them regularly to better understand their disease. The visits will include questions, a physical exam, blood drawing, a lumbar puncture, and a skin biopsy. The visits will also include tests that assess the electrical conductivity of the patients' nerves as well as a test to measure the patients' brain wave activity. In addition, the investigators will be performing tests to evaluate the patients' motor function, their vision, and thinking ability. Identifying an effective GAN treatment is very important because there is currently none. Clinical trials are the only way to decide whether a new treatment works in GAN patients or not.

With the future objective of conducting clinical trials in GAN, the proposed project has three specific aims. The first is to plan for clinical trials by developing reliable outcome measures, and establishing the infrastructure needed to carry out efficient clinical trials. The second is to further characterize the patient population from a clinical and molecular point of view, and the third aim is to utilize the information gathered in this study to further pre-clinical GAN drug development to select candidate drugs.

DETAILED DESCRIPTION:
Giant Axonal Neuropathy (GAN) is a rare autosomal recessive neurodegenerative disorder that appears during childhood and affects both the central and peripheral nervous systems. This disorder is generally characterized by motor and sensory involvement including progressive and predominant distal clumsiness, muscle weakness, and pronounced gait disturbances. GAN is caused by various mutations in the GAN gene that encodes the protein gigaxonin. This leads to giant axonal swelling and degeneration due to substantial accumulation of neurofilaments in the axon. Currently, there is no effective therapy, with onset occurring before the age of seven, and death usually occurring between the first and third decade of life.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of Giant Axonal Neuropathy.
2. Documentation of the presence of a mutation in the GAN gene as determined by gene sequencing from a CAP/CLIA certified laboratory or an equivalent organization.
3. Parents or if applicable subjects must give informed consent must be capable of complying with the study procedures.
4. Willing and able to comply with all protocol requirements and procedures.

Exclusion Criteria:

1. Unwilling or unable to travel to Columbia University Medical Center.
2. Unstable medical condition precluding participation.
3. Significant respiratory compromise that would interfere with safe travel to site of evaluation.
4. Having a contraindication to the MRI safety requirements, including pacemaker or other implanted electrical device, brain stimulator, some types of dental implants, aneurysm clips (metal clips on the wall of a large artery), metallic prostheses (including metal pins and rods, heart valves, and cochlear implants), implanted delivery pump, shrapnel fragments, or history of claustrophobia.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: People diagnosed with Giant Axonal Neuropathy
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2011-12; Primary Completion 2014-12 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Gross Motor Function Measure (GMFM) | Up to 24 months

SECONDARY OUTCOMES:
Nerve Conduction Study (NCS)/Motor Unit Number Estimation (MUNE) | Up to 24 months
Somatosensory Evoked Potential (SSEP) | Up to 24 months
Brainstem Auditory Evoked Response (BAER) | Up to 24 months
Pulmonary Function Testing (PFT)/Forced Vital Capacity (FVC) | Up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Darryl DeVivo, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Pediatric Neuromuscular Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — http://hannahshopefund.org/